CLINICAL TRIAL: NCT06921889
Title: Investigating the Biomechanical and Functional Outcomes of Autologous Chondrocyte Implantation: A Multi-centre Study
Brief Title: The Biomechanical Outcomes of Autologous Chondrocyte Implantation
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Gwenllian Tawy, Dr, University of Manchester
Other Study IDs: v1 04/08/2023
Record Dates: First submitted 2025-03-24; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chondral Defect
Keywords: Chondral defect; Cartilage repair; Knee; Autologous chondrocyte implantation; Biomechanical outcome; Gait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Participant: All participants of this study will be undergoing an autologous chondrocyte implantation of the knee for a chondral defect.
  Interventions: Procedure: Autologous Chondrocyte Implantation (ACI)

INTERVENTIONS:
Procedure: Autologous Chondrocyte Implantation (ACI) — ACI is a two-stage process that utilises the patient's own chondrocytes to repair damaged chondral tissue. After a harvesting procedure to obtain the cells, the chondrocytes are cultured and expanded in a specialised laboratory. A second procedure is then performed to implant the cells into the defect to replace and regenerate the injured cartilage. ACI allows the knee to generate durable and hyaline-like repair tissue.

SUMMARY:
Injury to the knee can damage the lining of the knee's bones, called cartilage. Cartilage injuries cause pain and limit movement, making activities like walking, playing sports, and working difficult.

Cartilage cannot repair itself well, so surgery is often needed to repair it. People who have cartilage repair surgery want to return to normal activities after their operation. Doctors and scientists know the operation can reduce pain, but do not fully understand how it affects movement.

This research will help us see if knee function gets better after cartilage repair surgery. The results will help doctors and patients understand what to expect from the surgery. It could also uncover common problems after surgery that could be fixed with physiotherapy.

This research is important because untreated cartilage injuries can develop into arthritis later in life. Arthritis is a painful lifelong condition that could be prevented by effectively treating the cartilage injury.

In this study, adult patients who are waiting to have a type of cartilage repair surgery called 'autologous chondrocyte implantation' (ACI) at one of 7 hospitals will be invited to take part in the study by their surgeon. Patients who decide to take part will be invited to two appointments at their own hospital, where assessments of their knee function will be performed. The tests will assess the knee's movement, and the patient's balance and walking abilities. The first research appointment will take place before the operation, and the second and final appointment will take place 6-months after surgery. The results of this study will help us understand how knee function changes after cartilage repair surgery.

The study will take place across 7 ACI centres in England, and is funded by Orthopaedic Research UK and the British Association for Surgery of the Knee.

DETAILED DESCRIPTION:
Knee joint articular cartilage is a primary load-bearing surface that endures repetitive high impact loading during activities of daily living. Individuals of any age can injure the knee's articular cartilage. However, as cartilage has an innate limited capacity to regenerate, surgical interventions that adopt tissue engineering techniques are often necessary to repair cartilage and preserve the joint.

Autologous chondrocyte implantation (ACI) is a surgical procedure that is offered to some patients with focal cartilage injuries of the knee. The first pilot study on the use of ACI in humans was published by Brittberg and colleagues in 1994. By 2010 35,000 ACI procedures had been performed worldwide.

Patient-reported outcomes and survivorship of ACI have been well reported in current literature. However, objective biomechanical and functional outcomes of ACI patients are not well understood. This knowledge is essential for optimising treatment, because poor functional outcome is known to worsen quality of life. This is particularly true for patients of working age who wish to return to an active and independent lifestyle.

The applicant recently conducted and published a systematic review on the functional outcome of ACI. The review identified only 19 eligible articles of 20 ACI cohorts. The data showed that the average range of motion (ROM) improved with clinical (>5˚) and statistical significance (p < 0.05) postoperatively: 130.5± 14.8˚ to 136.1±10.2º, however only 7 studies reported both pre- and post-operative RoM. Knee strength significantly improved within the first two postoperative years but remained poorer than control groups at final follow-up (n=11). The review also found no statistical differences between ACI and control groups in their ability to perform functional activities like the 6-minute walk and hop tests post-operatively (n = 8). Only two papers had published on the kinematics of gait post-operatively. Both papers reported the outcomes of the same cohort, stating that there were no significant differences in spatio-temporal parameters between ACI patients and controls post-operatively. However, kinematic differences were observed during two specific phases of the gait cycle. Differences were also reported in peak knee adduction and peak knee extension moments.

The limited literature identified by this review highlighted the urgent need for research into the functional outcomes of joint preservation surgeries like ACI to optimise functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chondral injury to the knee by a consultant orthopaedic surgeon Participants must have this diagnosis, else they are not eligible for ACI surgery.
* Listed for ACI for a chondral injury by a consultant orthopaedic surgeon Participants must be listed for ACI, as this is the treatment of interest in this research study
* Over 18 years old Participants must be legally capable of providing informed consent for the study.

Exclusion Criteria:

* Listed for any treatment other than ACI Participants must be listed for ACI, as this is the treatment of interest in this research study
* Under 18 years old. Participants must be legally capable of providing informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing ACI surgery for a chondral lesion in the knee.
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Knee range of motion measured in degrees with a goniometer | 6 months
  Change in knee range of motion in degrees post-operatively.

SECONDARY OUTCOMES:
Gait kinematics measured by motion capture technology | 6 months
  Changes to gait kinematics (angles in degrees) post-operatively
Gait kinetics measured by motion capture technology | 6 months
  Changes to gait kinetics (force in Newton) post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Gwenllian F Tawy, PhD, Principal Investigator — University of Manchester
Locations (7):
- United Kingdom (7):
  - Royal Orthopaedic Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Chapel Allerton Orthopaedic Centre, Leeds
  - Trafford General Hospital, Manchester
  - Southampton General Hospital, Southampton
  - Royal National Orthopaedic Hospital, Stanmore
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
No identifiable information will be published from this research. Only anonymised data will be shared to the public.